CLINICAL TRIAL: NCT04925505
Title: Usefulness of Pulse Oximeter Perfusion Index for Predicting the Success of Interscalene Brachial Plexus Blockade Under General Anesthesia
Brief Title: Perfusion Index for Predicting Brachial Plexus Block Success Under General Anesthesia
Status: Completed | Type: Observational
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Seok Kyeong Oh, Assistant professor, Korea University Guro Hospital
Other Study IDs: 2021GR0104
Record Dates: First submitted 2021-06-02; First posted 2021-06-14 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Disorder of Shoulder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BPB success: The study included patients aged between 20 and 70 yr who are to undergo elective shoulder surgery under general anesthesia. Patients undergo general anesthesia induction before the interscalene block is performed. Ultrasound-guided interscalene brachial plexus block will be performed in anesthetized patients before surgery. PI monitor will be applied to both blocked and non-blocked limbs using two separate oximeters. And the SUCCESS (or failure) of the block will be confirmed by (1) 30% change of heart rate and blood pressure after incision during operation, and (2) pain score, motor and sensory function test after surgery in the post-anesthesia recovery unit.
  Interventions: Procedure: Interscalene brachial plexus blocks with ultrasound guidance under general anesthesia
- BPB failure: The study included patients aged between 20 and 70 yr who are to undergo elective shoulder surgery under general anesthesia. Patients undergo general anesthesia induction before the interscalene block is performed. Ultrasound-guided interscalene brachial plexus block will be performed in anesthetized patients before surgery. PI monitor will be applied to both blocked and non-blocked limbs using two separate oximeters. And the (success or) FAILURE of the block will be confirmed by (1) 30% change of heart rate and blood pressure after incision during operation, and (2) pain score, motor and sensory function test after surgery in the post-anesthesia recovery unit.
  Interventions: Procedure: Interscalene brachial plexus blocks with ultrasound guidance under general anesthesia

INTERVENTIONS:
Procedure: Interscalene brachial plexus blocks with ultrasound guidance under general anesthesia — Ultrasound-guidance, interscalene brachial plexus blocks, in-plane technique, perineural injection, 0.5% ropivacaine 12.5ml and 0.2% lidocaine 12.5ml

SUMMARY:
This study was designed to determine whether the success or failure of interscalene brachial plexus block under general anesthesia can be predicted using perfusion index (PI).

DETAILED DESCRIPTION:
The success of peripheral nerve blocks is usually evaluated by assessment of sensory and motor function; however, this method cannot be applied in the patient who has uncheckable mental status, e.g. general anesthesia, or who is uncommunicable, e.g. different language user.

The perfusion index (PI) is a numerical value for the ratio between pulsatile and non-pulsatile blood flow measured by a special pulse oximeter, and PI had been proved as a useful tool for evaluation of successful supraclavicular nerve block in awake patients as an objective method.

With the use of ultrasound guidance in skilled hands, it is a reasonable option to perform neuraxial and peripheral regional blocks in sedated or anesthetized patients. However, there has been no evidence of applying PI for predicting the success of nerve block in general anesthetized patients.

ELIGIBILITY:
Inclusion Criteria:

* 20-70 years old,
* BMI 20-35 kg.m-2,
* elective shoulder surgery,
* ASA physical status I-III

Exclusion Criteria:

* refusal of the patient,
* comorbid with serious vascular disease,
* diabetes,
* allergy to local anesthetics,
* patients on regular opioids,
* peripheral neuropathy.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients aged 20-70 who are scheduled for shoulder surgery under general anesthesia, with ASA physical status I-III
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Perfusion Index | change between before and 15 minutes after brachial plexus block
  perfusion index measured applied to both blocked and non-blocked limbs using two separate oximeters

SECONDARY OUTCOMES:
Heart rate | change between before and 5 minutes after incision of surgical procedure
  heart rate in bpm during operation
Blood pressure | change between before and 5 minutes after incision of surgical procedure
  blood pressure in mmHg during operation
Pain score | 1 hour after surgery
  Numeric rating scale for pain on a 0-10 scale where 0=no pain and 10=unbearable pain
Sensory function test on supraclavicular nerve and axillary nerve | 1 hour after surgery
  0-2 scale where 0=no block; 1=analgesia (patient can feel touch, not cold); 2=anesthesia (patient cannot feel touch)
Motor function test on supraclavicular nerve and axillary nerve and | 1 hour after surgery
  0-2 scale where 0 = no block; 1 = paresis; 2 = paralysis

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abdelnasser A, Abdelhamid B, Elsonbaty A, Hasanin A, Rady A. Predicting successful supraclavicular brachial plexus block using pulse oximeter perfusion index. Br J Anaesth. 2017 Aug 1;119(2):276-280. doi: 10.1093/bja/aex166. PMID 28854539
- [Background] Misamore G, Webb B, McMurray S, Sallay P. A prospective analysis of interscalene brachial plexus blocks performed under general anesthesia. J Shoulder Elbow Surg. 2011 Mar;20(2):308-14. doi: 10.1016/j.jse.2010.04.043. Epub 2010 Aug 13. PMID 20708419
- [Background] Marhofer P. Regional blocks carried out during general anesthesia or deep sedation: myths and facts. Curr Opin Anaesthesiol. 2017 Oct;30(5):621-626. doi: 10.1097/ACO.0000000000000504. PMID 28696947